CLINICAL TRIAL: NCT04865419
Title: A Modular Phase I/II, Open-Label, Multi-Centre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AZD0466 Monotherapy or in Combination in Patients With Advanced Haematological Malignancies
Brief Title: Study of AZD0466 Monotherapy or in Combination in Patients With Advanced Haematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial terminated based on benefit-risk profile assessment
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8241C00001; 2020-005106-25 (EudraCT Number)
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Haematological Malignancies
Keywords: Pharmacokinetics; AZD0466; Voriconazole; Drug-drug interaction
MeSH Terms: interventions — AZD0466; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1: AZD0466 monotherapy (Experimental): Participants will receive intravenous infusion of AZD0466 monotherapy once weekly during Cycle 1 (35 days), Cycle 2 (28 days) and Cycle 3 (28 days) and also beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: AZD0466
- Module 2: AZD0466 + Voriconazole (Experimental): Participants may receive IV infusion of AZD0466 in combination with or without voriconazole during Cycle 1 (21 days), and Cycle 2 (28 days) and Cycle 3 (28 days) and also beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: AZD0466; Drug: Voriconazole

INTERVENTIONS:
Drug: AZD0466 — AZD0466 powder for concentrate for solution for infusion will be administered by IV infusion.
Drug: Voriconazole — Voriconazole film-coated tablet will be administered orally.
  Arms: Module 2: AZD0466 + Voriconazole

SUMMARY:
The purpose of the study is to the evaluate safety, tolerability, pharmacokinetics (PK), and efficacy of AZD0466 as monotherapy in partciapants with advanced haematological malignancies and also to assess drug-drug interaction (DDI) potential between AZD0466 and the azole antifungal voriconazole.

DETAILED DESCRIPTION:
The study consists of 2 individual modules as: Module 1 (AZD0466 monotherapy), and Module 2 (DDI study of AZD0466 with voriconazole).

Eligible participants will be assigned to study treatments across Modules 1 and 2.

1. Module 1: AZD0466 monotherapy will include 2 parts- Part A dose escalation cohorts and Part B dose expansion cohorts. Initiation of Part B will depend on the evaluation of safety, tolerability, and PK in Part A.
2. Module 2: AZD0466 and voriconazole DDI study.

All participants will receive AZD0466, and administration will continue until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukaemia (AML) or acute lymphoblastic leukaemia (ALL), or intermediate or higher risk myelodysplastic syndrome (MDS; Part A only), which is histologically proven based on criteria established by the World Health Organization (WHO) as documented by medical records. for which there are limited treatment options known to provide clinical benefit.
* Eastern cooperative oncology group performance status ≤2. Performance status must not have deteriorated by ≥2 levels within 2 weeks after providing informed consent.
* Predicted life expectancy ≥8 weeks.
* Adequate organ function at screening as per the protocol defined criteria.
* Adequate cardiac function as demonstrated by LVEF > 50% on screening cardiac multigated acquisition, magnetic resonance image or echocardiogram.
* Willing and able to participate in all required study evaluations and procedures including receiving IV administration of study treatment and admission to the hospital, when required, for administration of study treatment and monitoring.
* For inclusion in the genetic component of the study, participants must fulfil protocol defined criteria.
* White blood cell count must be <10 x 10^9/L prior to the first dose in Cycle 1, Day 1. Treatment with hydroxyurea during screening and Cycle 1 to control white blood cell count is permitted.
* Women of childbearing potential and men should use protocol defined contraceptive measures.

Exclusion Criteria:

* Unresolved toxicity from prior anticancer therapy of Common Terminology Criteria for Adverse Events Grade ≥2. Participants with Grade 2 neuropathy or Grade 2 alopecia are eligible.
* Active idiopathic thrombocytopenic purpura.
* Stem cell transplant < 100 days prior to the first dose of study treatment.
* Immunosuppression for graft versus host disease (GVHD) or GVHD prophylaxis within 4 weeks prior to the first dose of study treatment.
* Active central nervous system (CNS) leukaemia/leptomeningeal disease/spinal cord compression. Participants who have a history of CNS leukaemia must be free of CNS leukaemia for >30 days prior to the first dose of study treatment, and the most recent 2 lumbar punctures must be negative for leukaemic cells, to be eligible.
* Known uncontrolled infection with cytomegalovirus (CMV) infection (positive CMV Immunoglobulin M (IgM) and/or positive polymerase chain reaction (PCR) result).
* Active infection including human immunodeficiency virus, Hepatitis B, Hepatitis C, or severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2).
* As judged by the Investigator: any evidence of severe or uncontrolled systemic diseases, (eg, severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]); current unstable or uncompensated respiratory or cardiac conditions; Uncontrolled hypertension; history of, or active, bleeding diatheses (eg, haemophilia or von Willebrand disease); uncontrolled active systemic fungal, bacterial, or other infection.
* Any of the given cardiac criteria: history of myocarditis within one year of study entry, or heart failure New York Heart Association Functional Classification Class 3 or 4; mean resting corrected QT interval (QTcF) ≥470 msec obtained from 3 electrocardiogram (ECGs), in the absence of a cardiac pacemaker; abnormalities in rhythm, conduction or morphology of resting ECG; any factors that increase the risk of QTc prolongation or risk of arrhythmic events such congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age.
* History of another life-threatening malignancy ≤2 years prior to first dose of study treatment. The following are permitted: myelodysplastic syndrome or myeloproliferative neoplasm (including chronic myelomonocytic leukaemia [CMML]); malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening and considered to be at low risk of recurrence by the treating physician; adequately treated lentigo malignant melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer; adequately treated carcinoma in situ without current evidence of disease.
* Any of the mentioned procedures or conditions currently or in the 6 months prior to the first dose of study treatment: coronary artery bypass graft; angioplasty; vascular stent; myocardial infarction; angina pectoris; haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other CNS bleeding.
* Treatment with any of the mentioned therapy: radiotherapy less than 3 weeks prior to first study treatment; chemotherapy within ≤14 days or 5 half-lives prior to the first dose of study treatment. Treatment with high-dose steroids for primary malignancy control is permitted but must be discontinued at least 2 days prior to the first dose of study treatment. Treatment with hydroxyurea is permitted; immunotherapies and cellular therapies within 4 weeks prior to the first dose of study treatment; investigational drugs within ≤14 days or 5 half-lives (whichever is shorter) prior to the first dose of study treatment; major surgery (excluding placement of vascular access) ≤21 days, or minor surgical procedures ≤7 days, prior to the first dose of study treatment. No waiting is required mentioned implantable port or catheter placement; prescription or non-prescription drugs or other products known to be sensitive substrates of BCRP, OCT2, OAT3, OATP1B1, OATP1B3, CYP2B6, CYP2C8, CYP2C9 or CYP2D6, or reversible moderate or strong CYP3A inhibitors, which cannot be discontinued within 5 half-lives prior to the first dose of study treatment and withheld throughout the study until 14 days after the last dose of AZD0466; moderate or strong mechanism-based inhibitors or inducers of CYP3A4 which cannot be discontinued within 5 half-lives plus of the specific drug 12 days of the drug prior to the first dose of study treatment and withheld until 14 days after the last dose of AZD0466; concurrent anti-coagulation therapy, including aspirin and heparin, which cannot be stopped; medications with known risk of Torsades de Pointes which cannot be discontinued within 5 half-lives of the first dose of study treatment and withheld until 14 days after the last dose of AZD0466; IV anti infection treatment within 14 days before first dose of study treatment.
* History of hypersensitivity to polyethylene glycol (PEG), PEGylated products or drugs with a similar chemical structure or class to AZD0466 or other BH3 mimetic.

Module 2:

• Patients for whom treatment with voriconazole is contraindicated per the local prescribing information must not enter the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MD, PhD, Principal Investigator — The University of Texas MD Anderson Cancer Center 1515 Holcombe Boulevard, Unit 431 Houston, Texas 77030 United States of America
Locations (15):
- United States (5):
  - Research Site, Duarte, California
  - Research Site, Jacksonville, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Columbus, Ohio
  - Research Site, Houston, Texas
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Parkville
- Research Site, Pessac, France
- Germany (3):
  - Research Site, Aachen
  - Research Site, Heidelberg
  - Research Site, Kiel
- Italy (3):
  - Research Site, Bologna
  - Research Site, Meldola
  - Research Site, Rozzano
- Research Site, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8241C00001&attachmentIdentifier=93635c8f-d911-475c-83a1-2da0b28302f6&fileName=Final_to_Sponsor_CSP_Redacted_PDFA.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8241C00001&attachmentIdentifier=59624dad-6fbf-4eea-bed1-e81bdd2f7df9&fileName=Final_to_Sponsor_SAP_Redacted_PDFA.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8241C00001&attachmentIdentifier=ea5d335e-0a9e-46ea-b477-406492b799c5&fileName=Final_to_sponsor_CSR-synopsis-ERV_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 modules. Module 1 of the study was conducted at 14 sites in 6 countries (Australia, France, Germany, Italy, South Korea, and United States of America [USA]). Module 2 of the study was conducted at 6 sites in 2 countries (Australia and USA).
Pre-assignment Details: Participants who met all the inclusion and none of the exclusion criteria were enrolled in this study. All study assessments were performed as per the schedule of assessment.
Groups:
- Module 1: AZD0466 Monotherapy- 300 mg: Participants received intravenous (IV) infusion of AZD0466 monotherapy once weekly during Cycle 1 (35 days), Cycle 2 (28 days) and Cycle 3 (28 days) and also beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
- Module 1: AZD0466 Monotherapy- 600 mg; Module 1: AZD0466 Monotherapy- 1200 mg; Module 1: AZD0466 Monotherapy- 2400 mg; Module 1: AZD0466 Monotherapy- 3600 mg; Module 1: AZD0466 Monotherapy- 5400 mg: Participants received IV infusion of AZD0466 monotherapy once weekly during Cycle 1 (35 days), Cycle 2 (28 days) and Cycle 3 (28 days) and also beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
- Module 2: AZD0466 300 mg+ Voriconazole; Module 2: AZD0466 600 mg+ Voriconazole; Module 2: AZD0466 1200 mg+ Voriconazole; Module 2: AZD0466 2400 mg+ Voriconazole; Module 2: AZD0466 3600 mg+ Voriconazole: Participants received IV infusion of AZD0466 both with and without voriconazole in Cycle 1. Participants received AZD0466 alone from Cycle 2 (28 days) onwards and beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole
Started | 4 | 4 | 7 | 5 | 10 | 2 | 1 | 3 | 4 | 4 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 7 | 5 | 10 | 2 | 1 | 3 | 4 | 4 | 2
Not completed — Other | 1 | 2 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 3 | 1 | 4 | 2 | 5 | 2 | 1 | 1 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) which consisted of all enrolled participants who received at least 1 dose of AZD0466.
Groups:
- Module 1: AZD0466 Monotherapy- 300 mg; Module 1: AZD0466 Monotherapy- 600 mg; Module 1: AZD0466 Monotherapy- 1200 mg; Module 1: AZD0466 Monotherapy- 2400 mg; Module 1: AZD0466 Monotherapy- 3600 mg; Module 1: AZD0466 Monotherapy- 5400 mg: Participants received IV infusion of AZD0466 monotherapy once weekly during Cycle 1 (35 days), Cycle 2 (28 days) and Cycle 3 (28 days) and also beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole | Total
Number analyzed (Participants) | 4 | 4 | 7 | 5 | 10 | 2 | 1 | 3 | 4 | 4 | 2 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Two separate rows have been created for each module to present the total Mean and S.D. separately for each module as different population of participants were involved in each module.
  Years
    Module 1: number analyzed (Participants) | 4 | 4 | 7 | 5 | 10 | 2 | 0 | 0 | 0 | 0 | 0 | 32
    Module 1 | 61.3 (20.07) | 72.3 (4.03) | 64.6 (14.98) | 63.4 (16.91) | 62.8 (10.77) | 61.5 (10.61) |  |  |  |  |  | 64.2 (12.99)
    Module 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 4 | 2 | 14
    Module 2 |  |  |  |  |  |  | NA (NA) — Mean is not reported due to concerns with participant's confidentiality. Standard deviation is not calculable for 1 participant | 74.0 (5.20) | 40.0 (20.99) | 62.5 (17.08) | 71.0 (7.07) | 61.0 (19.89)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | NA — Data are not reported due to concerns with participant's confidentiality. | 2 | 3 | 3 | 5 | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Data are not reported due to concerns with participant's confidentiality. | 0 | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data are not reported due to concerns with participant's confidentiality. | 2 | 4 | 2 | 5 | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Data are not reported due to concerns with participant's confidentiality. | 3 | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Data are not reported due to concerns with participant's confidentiality. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 3 | 6 | 5 | 9 | 0 | 0 | 3 | 4 | 3 | 2 | 35
  Other | 3 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 9
  Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) [Module 1]
Description: The safety and tolerability of AZD0466 in participants with advanced haematological malignancies were assessed.
Time Frame: From screening (Day -28 to Day 1) up to 28 days after last dose (Approximately 2.1 years)
Population: Safety analysis set consisted of all enrolled participants who received at least 1 dose of AZD0466.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg
Number analyzed (Participants) | 4 | 4 | 7 | 5 | 10 | 2
Participants
  Any AE | 4 | 4 | 6 | 5 | 9 | 2
  Any SAE | 4 | 0 | 3 | 3 | 8 | 1
  Any SAE with outcome death | 0 | 0 | 0 | 0 | 1 | 0
  Any AE leading to discontinuation of AZD0466 | 0 | 0 | 0 | 0 | 3 | 1
  Any possibly related AE | 3 | 2 | 3 | 4 | 8 | 2
  Any possibly related SAE | 0 | 0 | 0 | 2 | 2 | 1
  Any AE leading to AZD0466 dose reduction | 0 | 0 | 0 | 0 | 0 | 1
  Any AE leading to AZD0466 dose interruption | 0 | 1 | 2 | 3 | 5 | 1
  Any AE of >= CTCAE grade 3 | 4 | 2 | 4 | 4 | 9 | 2
  Any SAE and/or >= CTCAE grade 3 AE | 4 | 2 | 4 | 4 | 9 | 2
  Any AE classified as a DLT | 0 | 0 | 0 | 0 | 2 | 1
  Any possibly related deaths | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) [Module 2]
Description: The safety and tolerability of AZD0466 in participants with advanced haematological malignancies were assessed.
Time Frame: From screening (Day -28 to Day 1) up to 28 days after last dose (Approximately 2.1 years)
Population: Safety analysis set consisted of all enrolled participants who received at least 1 dose of AZD0466.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole
Number analyzed (Participants) | 1 | 3 | 4 | 4 | 2
Participants
  Any AE | 1 | 3 | 3 | 4 | 2
  Any SAE | 1 | 2 | 0 | 4 | 2
  Any SAE with outcome death | 0 | 0 | 0 | 1 | 0
  Any AE leading to discontinuation of AZD0466 | 1 | 0 | 0 | 0 | 1
  Any possibly related AE | 1 | 1 | 2 | 3 | 2
  Any possibly related SAE | 0 | 0 | 0 | 2 | 1
  Any AE leading to AZD0466 dose reduction | 0 | 1 | 1 | 0 | 0
  Any AE leading to AZD0466 dose interruption | 0 | 2 | 1 | 1 | 2
  Any AE of >= CTCAE grade 3 | 1 | 3 | 3 | 4 | 2
  Any SAE and/or >= CTCAE grade 3 AE | 1 | 3 | 3 | 4 | 2
  Any AE classified as a DLT | 0 | 0 | 0 | 0 | 0
  Any possibly related deaths | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT) [Module 1]
Description: The safety and tolerability of AZD0466 in participants with advanced haematological malignancies were assessed.
Time Frame: upto 35 days
Population: DLT-evaluable set consisted of participants enrolled in the dose-escalation that have received at least 3 doses of AZD0466 at the target dose level (75% of target doses from Day 8 to Day 29 in Cycle 1) and have completed the safety follow-up through the DLT evaluation period or have experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 7 | 1
Participants | 0 | 0 | 0 | 0 | 2 | 1

4. Secondary Outcome: Module 1: Complete Response Rate
Description: Complete response rate (CR+CRi) is defined as the percentage of participants who have a complete remission (CR) or incomplete haematological response (CRi).
Time Frame: Day 1 until post treatment follow-up (28 days after last dose) (approximately 2.1 years)
Population: Intention to treat (ITT) set consisted of all enrolled participants who received at least 1 dose of AZD0466.
Measure: Number; unit: Percentage of participants
Groups:
- Module 1: AZD0466 Monotherapy- 300 mg- Acute Lymphoblastic Leukaemia (ALL); Module 1: AZD0466 Monotherapy- 1200 mg - ALL; Module 1: AZD0466 Monotherapy- 3600 mg- ALL: Participants received intravenous infusion of AZD0466 monotherapy once weekly during Cycle 1 (35 days), Cycle 2 (28 days) and Cycle 3 (28 days) and also beyond Cycle 3 until progressive disease, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg | Module 1: AZD0466 Monotherapy- 300 mg- Acute Lymphoblastic Leukaemia (ALL) | Module 1: AZD0466 Monotherapy- 1200 mg - ALL | Module 1: AZD0466 Monotherapy- 3600 mg- ALL
Number analyzed (Participants) | 2 | 4 | 6 | 5 | 8 | 2 | 2 | 1 | 2
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Module 1: Time to Response (TTR)
Description: Time to response is defined as the time from date of first dose until the date of first documented CR or CRi.
Time Frame: Day 1 until post treatment follow-up (28 days after last dose) (Approximately 2.1 years)
Population: ITT set consisted of all enrolled participants who received at least 1 dose of AZD0466.
  Since none of the participants had achieved CR or CRi, TTR could not be calculated.
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Module 1: Duration of Response
Description: Duration of Response (DoR) will be defined as the time from the date of first documented response (CR+CRi) until date of documented progression, relapse or failure or death due to any cause.
Time Frame: Day 1 until post treatment follow-up (28 days after last dose) (approximately 2.1 years)
Population: ITT set consisted of all enrolled participants who received at least 1 dose of AZD0466.
  Since none of the participants had achieved CR or CRi, DoR could not be calculated.
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Module 1: Overall Survival
Description: Overall survival (OS) is defined as time from date of first dose until the date of death due to any cause.
Time Frame: Day 1 until post treatment follow-up (28 days after last dose) and survival follow-up (every month after last dose) (approximately 2.1 years)
Population: ITT set consisted of all enrolled participants who received at least 1 dose of AZD0466.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg
Number analyzed (Participants) | 4 | 4 | 7 | 5 | 10 | 2
Months | 3.2 [2.7 to NA] — The value was not calculated due to low number of events | NA [1.3 to NA] — The value was not calculated due to low number of events | 3.8 [2.1 to NA] — The value was not calculated due to low number of events | NA [1.1 to NA] — The value was not calculated due to low number of events | 2.4 [0.5 to NA] — The value was not calculated due to low number of events | 2.0 [0.9 to NA] — The value was not calculated due to low number of events

8. Secondary Outcome: Module 2: Area Under the Plasma Concentration-curve (AUC) of AZD4320 After Administration of AZD0466 Alone and in Combination With Voriconazole
Description: Assessment of AUC to evaluate the drug-drug interaction potential between AZD0466 and the azole antifungal voriconazole.
  For this outcome measure, pharmacokinetics (PK) analysis set was included which consisted of all dosed participants with reportable plasma concentrations and no important AEs or protocol deviations that may affect PK.
Time Frame: Cycle 1 Days 1, 2, 3, 4, 8 and days 15, 16, 17, 18, 19, and Cycle 2 Day 1, Cycle 3 Day 1 and beyond (Cycle length 28-days) (approximately 2.1 years)
Population: It was pre-specified by the Study Protocol to only analyze dosed participants with at least 1 reportable plasma concentration and no important AEs or protocol deviations that may impact PK for this Outcome Measure.
  Due to changes in target dose levels and protocol deviations affecting derivation of PK parameters, AUC could not be statistically assessed (summary statistics or inferential statistical comparisons), as no participant met pre-specified criteria for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomole/liter (h*nmol/L)
Arm/Group | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole
Number analyzed (Participants) | 1 | 3 | 4 | 4 | 2
hours*nanomole/liter (h*nmol/L) | NA (NA) — AUC could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — AUC could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — AUC could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — AUC could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — AUC could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol.

9. Secondary Outcome: Module 2: Maximum Observed Plasma (Peak) Drug Concentration (Cmax) of AZD4320 After Administration of AZD0466 Alone and in Combination With Voriconazole
Description: Assessment of Cmax to evaluate the drug-drug interaction potential between AZD0466 and the azole antifungal voriconazole.
  For this outcome measure, PK analysis set was included which consisted of all dosed participants with reportable plasma concentrations and no important AEs or protocol deviations that may affect PK.
Time Frame: Cycle 1: Days 1, 2, 3, 4, 8 and days 15, 16, 17, 18, 19, and Cycle 2 Day 1, Cycle 3 Day 1 and beyond (Cycle length 28-days) (approximately 2.1 years)
Population: It was pre-specified by the Study Protocol to only analyze dosed participants with at least 1 reportable plasma concentration and no important AEs or protocol deviations that may impact PK for this Outcome Measure.
  Due to changes in target dose levels and protocol deviations affecting derivation of PK parameters, Cmax could not be statistically assessed (summary statistics or inferential statistical comparisons), as no participant met pre-specified criteria for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)/liter (L)
Arm/Group | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole
Number analyzed (Participants) | 1 | 3 | 4 | 4 | 2
nanomole (nmol)/liter (L) | NA (NA) — Cmax could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — Cmax could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — Cmax could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — Cmax could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol. | NA (NA) — Cmax could not be summarized because no participants met pre-specified analysis criteria due to changes in target dose levels and protocol deviations affecting PK parameter derivation as specified in the study protocol.

10. Secondary Outcome: Module 1 and Module 2: Plasma Concentration of AZD4320
Description: Assessment of AZD4320 to characterise the PK profile of AZD0466 following intravenous administration (via PK profiles of the active moiety AZD4320 in plasma).
Time Frame: Module 1: Cycle 1 Days 1-30 (Cycle length 21 days) to Cycle 3 Days 1-28, & beyond (Cycle length 28 days); Module 2: Cycle 1 Days 1-8, Days 15-19 (Cycle length 21 days), Cycle 2 Day 1, Cycle 3 Day 1 & beyond (Cycle length 28-days) (approximately 2.1 Years)
Population: PK set consisted of all dosed participants with reportable plasma concentrations and no important AEs or protocol deviations that may affect PK.
  For PK concentration and parameter data, if there were <3 values available at a time point or if the value was below the lower limit of quantification (BLQ), descriptive statistics were reported as 'Not calculable (NC)' or 'Not Available (NA)'.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole
Number analyzed (Participants) | 4 | 4 | 7 | 5 | 10 | 2 | 1 | 3 | 4 | 4 | 2
nanomolar (nM)
  Released AZD4320: Cycle 1/ Day 8: number analyzed (Participants) | 4 | 4 | 7 | 2 | 7 | 2 | 1 | 3 | 3 | 4 | 2
  Released AZD4320: Cycle 1/ Day 8 | 528.6 (178.7) | 1053 (61.18) | 1651 (179.8) | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. | 4117 (141.6) | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. | 326.9 (33.08) | 1440 (11.20) | 1745 (62.40) | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP.
  Released AZD4320: Cycle 2/ Day 1: number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 0
  Released AZD4320: Cycle 2/ Day 1 | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. |  | 1371 (98.40) | 1872 (196.0) | 4661 (83.61) |  |  |  |  | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. |
  Total AZD4320: Cycle 1 /Day 8: number analyzed (Participants) | 3 | 4 | 7 | 3 | 7 | 2 | 1 | 3 | 3 | 4 | 1
  Total AZD4320: Cycle 1 /Day 8 | 16220 (53.05) | 48910 (28.88) | 104700 (76.62) | 200400 (27.12) | 272800 (22.27) | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. | 36150 (14.97) | 84700 (34.72) | 186100 (44.69) | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP.
  Total AZD4320: Cycle 2/ Day 1: number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 0 | 0 | 1 | 0 | 2 | 0
  Total AZD4320: Cycle 2/ Day 1 | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. |  | 82070 (17.95) | 221400 (33.80) | 314500 (25.27) |  |  | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. |  | NA (NA) — Data were not reported due to presence of insufficient number of participants for analysis at that timepoint in accordance with the SAP. |

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to Day 1) up to 28 days after last dose (Approximately 2.1 years).
Arm/Group | Module 1: AZD0466 Monotherapy- 300 mg | Module 1: AZD0466 Monotherapy- 600 mg | Module 1: AZD0466 Monotherapy- 1200 mg | Module 1: AZD0466 Monotherapy- 2400 mg | Module 1: AZD0466 Monotherapy- 3600 mg | Module 1: AZD0466 Monotherapy- 5400 mg | Module 2: AZD0466 300 mg+ Voriconazole | Module 2: AZD0466 600 mg+ Voriconazole | Module 2: AZD0466 1200 mg+ Voriconazole | Module 2: AZD0466 2400 mg+ Voriconazole | Module 2: AZD0466 3600 mg+ Voriconazole
All-Cause Mortality (participants affected / at risk) | 3/4 | 1/4 | 4/7 | 2/5 | 5/10 | 2/2 | 1/1 | 1/3 | 2/4 | 2/4 | 1/2
Serious Adverse Events (participants affected / at risk) | 4/4 | 0/4 | 3/7 | 3/5 | 8/10 | 1/2 | 1/1 | 2/3 | 0/4 | 4/4 | 2/2
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 6/7 | 5/5 | 9/10 | 2/2 | 1/1 | 3/3 | 3/4 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Module 1: AZD0466 Monotherapy- 300 mg (N=4) | Module 1: AZD0466 Monotherapy- 600 mg (N=4) | Module 1: AZD0466 Monotherapy- 1200 mg (N=7) | Module 1: AZD0466 Monotherapy- 2400 mg (N=5) | Module 1: AZD0466 Monotherapy- 3600 mg (N=10) | Module 1: AZD0466 Monotherapy- 5400 mg (N=2) | Module 2: AZD0466 300 mg+ Voriconazole (N=1) | Module 2: AZD0466 600 mg+ Voriconazole (N=3) | Module 2: AZD0466 1200 mg+ Voriconazole (N=4) | Module 2: AZD0466 2400 mg+ Voriconazole (N=4) | Module 2: AZD0466 3600 mg+ Voriconazole (N=2)
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Module 1: AZD0466 Monotherapy- 300 mg (N=4) | Module 1: AZD0466 Monotherapy- 600 mg (N=4) | Module 1: AZD0466 Monotherapy- 1200 mg (N=7) | Module 1: AZD0466 Monotherapy- 2400 mg (N=5) | Module 1: AZD0466 Monotherapy- 3600 mg (N=10) | Module 1: AZD0466 Monotherapy- 5400 mg (N=2) | Module 2: AZD0466 300 mg+ Voriconazole (N=1) | Module 2: AZD0466 600 mg+ Voriconazole (N=3) | Module 2: AZD0466 1200 mg+ Voriconazole (N=4) | Module 2: AZD0466 2400 mg+ Voriconazole (N=4) | Module 2: AZD0466 3600 mg+ Voriconazole (N=2)
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 1 | 5 | 1 | 0 | 0 | 1 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 3 | 1 | 0 | 2 | 1 | 2 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 3 | 2 | 1 | 0 | 0 | 2 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 2 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coagulation test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT shortened (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 2 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell sedimentation rate (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Citrobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Trial terminated based on benefit-risk profile assessment. Due to early termination of the study, Module 1 Part A and Module 2 were conducted, Module 1 Part B was not started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT04865419/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT04865419/SAP_001.pdf